CLINICAL TRIAL: NCT05506085
Title: Deep Brain Stimulation for Laryngeal Dystonia: From Mechanism to Optimal Application
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Rita R. Patel, Associate Professor, Speech & Hearing Sciences, Indiana University
Other Study IDs: 14578
Record Dates: First submitted 2022-07-19; First posted 2022-08-18 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Laryngeal Dystonia; Adductor Spastic Dysphonia of Dystonia
Keywords: deep brain stimulation
MeSH Terms: conditions — Dysphonia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Deep Brain Stimulation: Voice outcomes and Magnetic resonance imaging will be compared pre- and post-DBS (Deep brain stimulation) in patients with laryngeal dystonia and adductor laryngeal dystonia. The evaluators will be masked for analyzing the voice outcomes pre-and post-DBS
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Deep Brain Stimulation of Globus Pallidus interna

SUMMARY:
Deep Brain Stimulation (DBS) is a neurosurgical procedure used to treat tremors, and dystonia. This study will enroll people who have a form of focal dystonia that affects their vocal cords called Adductor Laryngeal dystonia (ADLD). Participants will undergo Deep Brain Stimulation surgery to treat laryngeal dystonia as part of their clinical care. Before surgery, as part of the study they will have specialized testing to study the movement of the vocal cords, as well as functional magnetic resonance imaging (fMRI). While in the operating room, researchers will examine brain waves to better understand how faulty brain firing patterns lead to dystonia. After surgery, and activation of the deep brain stimulator, participants will repeat speech testing and vocal cord imaging as well as magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ADLD and ADLD plus tremor, as diagnosed by routine clinical examination by laryngologist, speech language pathologist, and neurologist.
* Patients undergoing globus pallidus interna (GPi) deep brain stimulation (DBS) for ADLD with tremor
* Age range of 18-80 years
* Native speakers of American English will be recruited since there are known differences in voice and neural signals of native and non-native speakers
* No evidence for dementia as assessed by neurologist.
* No evidence for severe untreated mood disorder as assessed by neurologist, or as evident on self-report (Beck Depression Inventory-II score > 29, Beck Anxiety Inventory Score > 26.
* At least 3 months since last botulinum toxin injection and the patients would need to be fully symptomatic with no residual effects of botulinum toxin on voice quality.

Exclusion Criteria:

* Individuals younger than 18 years and older than 80 years of age.
* Women who plan to become pregnant during the study period or are currently breastfeeding.
* Prior history of stroke, brain surgery, or other neurological disorder besides the one under study.
* Prior laryngeal framework surgeries or other disorders affecting the vocal folds
* Patients who are asymptomatic due to treatment with botulinum toxin into the vocal folds.
* Presence of ferromagnetic implants and cardiac implants that would be contraindicated to MRI
* Gagging or discomfort that would preclude the placement of the endoscope to visualize the larynx
* Dementia, severe depression or severe anxiety.
* Any clinical condition or medication judged by the investigators to potentially preclude the patient from safely completing awake brain surgery and research protocols.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals presenting for routine neurology clinic appointments will be screened for clinical DBS (Deep brain stimulation) candidacy
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2030-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in total number of Vocal fold movements | Before surgery, within 24 hours after surgery, 6 -9 months after surgery
  Vocal fold movements will be quantified (vibratory breaks + micromotions+ aperiodicities) using high-speed videoendoscopy (HSV) on sustained phonation of the vowel, words, and sentence production. The videoendoscopic recording will be obtained
Change in Acoustic voice recordings | Before surgery, within 24 hours after surgery, 6-9 months after surgery
  Acoustic voice recordings will be obtained using a microphone. Acoustic measurement of voice (voicing percentage) will be obtained from sustained phonation of the vowel /a/, sentences and reading a paragraph.
Microelectrode recording | during surgery
  Microelectrode recording is performed routinely during DBS (Deep brain stimulation) surgery. The study procedure will be to record voice simultaneously on sustained phonation of the vowels, syllables, and sentences using the data acquisition system NI USM 6221 with a microphone and high-speed videoendoscopy. Beta and theta band power spectral density will be analyzed as measurements.

SECONDARY OUTCOMES:
Change in Neuropsychological testing: Trails A | Before surgery, and 6-9 months after surgery
  Neuropsychological testing will be obtained pre (standard of care for DBS surgery) and 6 months post DBS surgery (experimental) to evaluate psychomotor speed
Change in Neuropsychological testin: Trails B | Before surgery, and 6-9 months after surgery
  Neuropsychological testing will be obtained pre (standard of care for DBS surgery) and 6 months post DBS surgery (experimental) to evaluate mental flexibility
Change in Neuropsychological testing: Controlled Oral Word Association Animal fluency | Before surgery, and 6-9 months after surgery
  Neuropsychological testing will be obtained pre (standard of care for DBS surgery) and 6-9 months post DBS surgery (experimental) to evaluate verbal fluency
Change in Resting state Functional Magnetic Resonance Imaging (fMRI) | before surgery and 6-9 months after surgery
  Resting state Functional Magnetic Resonance Imaging (rs-FMRI)
Change in Voice Handicap Index | before surgery and 6-9 months after surgery
  A 30-point questionnaire to describe the voice and the effects of voice on their daily lives. The scores range from 0 to 120. 0 to 30 is a low score with minimal handicap and 61 to 120 is considered severe handicap, 31 to 60 moderate handicap
Change in Speech Intelligibility | before surgery and 6-9 months after surgery
  will be computed from the 2nd, 3rd, and 4th sentences of the Rainbow passage as the number of correct words identified.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Patel, PhD, Principal Investigator — Indiana University; S. Elizabeth Zauber, MD, Principal Investigator — Indiana University; Kunal Gupta, MD, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data from individual patient data (IPD) will be made available to other researchers on request. We also plan to post IPD after study completion on IUScholarWorks where other researchers could access it.